CLINICAL TRIAL: NCT01823458
Title: Evaluation of Behavioral Economics Patient Incentive Strategies for Health Management
Brief Title: Behavioral Economics Incentives for Health Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC4 AG039115 - 03; RC4AG039115 (NIH)
Record Dates: First submitted 2013-03-05; First posted 2013-04-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: behavioral economics; incentives; health behavior; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lottery Insurance (Experimental): All participants receive a one time, $10 payment for attending the first exercise class of the 12 week session. Participants in the 'Lottery Insurance' arm receive a lottery ticket valued at $20 for attending either a Monday or Tuesday exercise class. They have the option to insure their lottery ticket by attending a second exercise class during the week on either Wednesday or Thursday. If they do not attend the second class, they have a 90% chance of winning the weekly lottery. This sequence is repeated each week over the 12 week exercise session.
  Interventions: Behavioral: Lottery Insurance
- Standard Lottery (Experimental): All participants receive a one time, $10 payment for attending the first exercise class of the 12 week session. Subjects in the 'Standard Lottery' arm receive a lottery ticket valued at $20 for attending either a Monday or Tuesday exercise class. They also receive the expected value of the insurance ($2) for attending a second exercise class during the week on either Wednesday or Thursday. They have a 90% chance of winning the weekly lottery. This sequence is repeated each week over the 12 week exercise session.
  Interventions: Behavioral: Standard Lottery

INTERVENTIONS:
Behavioral: Lottery Insurance
  Arms: Lottery Insurance
Behavioral: Standard Lottery
  Arms: Standard Lottery

SUMMARY:
Incentives are increasingly being used to motivate health behavior in medical studies. Small cash payments conditional on certain health and welfare promoting behaviors have shown efficacy in both real world and experimental settings. Furthermore, in incentive studies, behavioral economics has been shown to amplify behavior change beyond what is possible with simple cash payments, but little is known about how varying incentive payment design may impact health behavior. The goal of the present study is to evaluate a new incentive payment instrument, lottery insurance, to determine its impact on adherence to the target health behavior, attendance at free exercise classes provided by QueensCare Family Clinics, a safety-net medical clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age
* BMI between 25-40
* Receiving care in QueensCare Family Clinics

Exclusion Criteria:

* Failure to obtain exercise clearance from physician

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Attendance at exercise classes | 12 weeks
  Attendance at exercise classes over the 12 week session will be analyzed across 'Lottery Insurance' and 'Standard Lottery' arms.

SECONDARY OUTCOMES:
Body Mass Index | Change from Baseline Body Mass Index at 12 weeks
  Change from Baseline Body Mass Index (based on Centers for Disease Control calculations) at 12 weeks (post exercise session) will be assessed.
HbA1c | Change from Baseline HbA1c at 12 weeks
  Change from Baseline glycemic control (measured as percentage glycosylated hemoglobin [HbA1c] as part of a fasting blood sample) at 12 weeks (post exercise session) will be assessed.
Blood Pressure | Change from Baseline Blood Pressure at 12 weeks
  Change from Baseline Blood Pressure at 12 weeks (post exercise session) will be assessed.
LDL cholesterol | Change from Baseline LDL at 12 weeks
  Change from Baseline LDL cholesterol (measured as part of a lipid panel) at 12 weeks (post exercise session) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Doctor, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- QueensCare Family Clinics, Los Angeles, California, United States